CLINICAL TRIAL: NCT04204538
Title: Evaluation of Dietary Practices and Assessment of Nutritional Status and Associated Risk Factors for Metabolic Syndrome in the Young Adult Population of Rwanda
Brief Title: Dietary Practices and Metabolic Syndrome in the Young Adult Population of Rwanda
Acronym: NutriTransit
Status: Completed | Type: Observational
Sponsor: University Ghent (Other)
Collaborators: University of Rwanda (Other); Institut de Recherche en Sciences de la Sante, Burkina Faso (Other Government)
Responsible Party: Sponsor
Other Study IDs: EC/2019/1577
Record Dates: First submitted 2019-11-27; First posted 2019-12-19 (Actual); Last update posted 2024-02-07 (Actual); Status verified 2024-02

CONDITIONS: Metabolic Syndrome; Nutritional Status; Diet Habit
Keywords: Food Frequency Questionnaire; Dietary patterns; Risk factors; metabolic syndrome; Nutritional transition
MeSH Terms: conditions — Metabolic Syndrome; Feeding Behavior

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Serum samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Urban: Young adults living in urban communities of Rwanda
  Interventions: Other: Dietary habits; Other: Risk factors associated with metabolic syndrome
- Rural: Young adults living in rural communities of Rwanda
  Interventions: Other: Dietary habits; Other: Risk factors associated with metabolic syndrome

INTERVENTIONS:
Other: Dietary habits — Data collected using food frequency questionnaire
Other: Risk factors associated with metabolic syndrome — Data collected on nutritional status, biochemical indicators and other risk factors associated with metabolic syndrome

SUMMARY:
Policy makers in Rwanda have recently highlighted the importance of promoting healthy diets and lifestyle in response to rapidly increasing rates of obesity. This project will provide evidence on shifts in diet and nutritional status in urban dwellers as compared to the traditional diet and lifestyle in rural areas as a basis for a targeted public health policy for Rwanda.

DETAILED DESCRIPTION:
Adequate diet has been known for many years to be a major lever to significantly decrease the risk for non-communicable diseases (NCD). However, mainly due to urbanization and improved economic status in low and middle income countries (LMICs), the traditional largely plant-based diets are being replaced by more energy-dense and nutrient poor diets, incorporating more animal foods and processed foods and fat, and with a decrease in consumption of fruits and vegetables and other plant based foods. This diet change together with a sedentary lifestyle are typical phenomena in LMICs that are driving the so-called nutrition transition that is typically accompanied by an increase in obesity and in NCD like metabolic syndrome, diabetes, cardiovascular diseases and cancer. In Rwanda, NCD lead to 36% of total deaths. Cancers, diabetes, cardiovascular diseases, and chronic respiratory diseases account for 82% of NCD deaths. The major risk factor is the raised blood pressure (34.4%) and the probability of dying between ages 30 and 70 years from those four main NCD is estimated to 19%.

The Government of Rwanda has installed an operational NCD unit in the Ministry of Health with a view to developing preventive strategies vis-à-vis the nutrition transition process in the country. It has been shown already that there is a need for adopting dietary behaviour change to prevent the epidemic of chronic diseases.

The aim of this PhD work is to contribute in generating evidence needed to develop targeted prevention strategies for NCD in a broader framework of informed health policy making in Rwanda.

Specific objectives:

1. To identify the changes in eating habits of different socio- economic subgroups in adults living in Kigali, in comparison to their peers in rural areas;
2. To assess nutritional status and body composition using several methods (BMI, skinfold thicknesses, sitting height and body build, fat and fat free mass), with the ultimate objective to establish population-body composition-derived BMI cut-offs for overweight and obesity in this population;
3. To assess and compare the prevalence of common risk factors for non-communicable disease (high BMI, low fruit and vegetable consumption, low physical activity and high blood pressure) between rural and urban areas;
4. To evaluate people's nutrition knowledge, aptitude and capacity (KAP), perception of obesity and normal weight and food insecurity levels as risks factors for adherence to healthy dietary practices and life style;
5. To generate information to be used by governments to improve dietary habits and physical activity through targeted interventions.

The data collected in a cross sectional study design. Validated questionnaires will be used to get information on socio-economic characteristics, dietary practices, physical activity, other lifestyle factors and psycho-social and emotional indicators.

ELIGIBILITY:
Inclusion Criteria:

* Permanent residence of the selected urban or rural villages
* Holding a valid health insurance card
* Aged between 18 and 35 years
* Signing informed consent form
* Registration in city demographic system, since study participants will be selected from population registration cards at village level,
* Accept enumerators for home visit and data collection
* Accept to visit the laboratory for blood sample collection,
* Not suffering from any chronic disease such as VIH/ AIDS, diabetes, asthma, etc.

Exclusion Criteria:

* Lactating, pregnant, and recently delivering (less than six month-postpartum) women
* Physical disabilities that can prevent participants from working
* Mental disability such as clinically diagnosed depression, anxiety disorders, eating disorders and addictive behaviors.

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Participants will be selected randomly from the general population. Eligible subjects who agree to participate (informed consent) will be enrolled in the study.
Sampling Method: Non-Probability Sample
Enrollment: 1247 (Actual)
Dates: Start 2021-11-01 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Prevalence of the different dietary patterns | Through study completion (an average of 6 months)
  Dietary patterns will be identified using exploratory factor analysis on the food groups collected using the semi-quantitative Food Frequency Questionnaire. The dietary pattern identified will differ from plant_based diet and legume_based diet to western diet.
Prevalence of large waist circumference | Through study completion (an average of 6 months)
  Large waist circumference [> 89 centimeters for women and >102 centimeters for men]
Prevalence of high triglyceride concentrations | Through study completion (an average of 6 months)
  High triglyceride level [>150 milligrams per deciliter (mg/dL)]
Prevalence of high-density lipoprotein (HDL) cholesterol | Through study completion (an average of 6 months)
  Reduced high-density lipoprotein (HDL) cholesterol [< 40 mg/dL in men or < 50 mg/dL in women]
Prevalence of high blood pressure | Through study completion (an average of 6 months)
  Increased blood pressure [> 130/85 mm Hg]
Prevalence of high levels of fasting blood sugar | Through study completion (an average of 6 months)
  Elevated fasting blood sugar [>100 mg/dL]
Prevalence of participants with nutrition knowledge | Through study completion (an average of 6 months)
  Nutritional knowledge of macronutrients, micronutrients, water intake, diet and disease will be collected using a multiple choice answers. Each question had one mark for every correct response chosen. Using a marking scheme for nutritional knowledge test the scores were rated on score percentages using eight cut off points, with scores less than 20% indicating a bad nutritional knowledge, 50-59% satisfactory and Excellent for those scoring 80% and more.

SECONDARY OUTCOMES:
Prevalence of Food Insecure Households | Through study completion (an average of 6 months)
  The Household Food Insecurity Access (HFIA) Score is a continuous measure of the degree of food insecurity in the household and is based on a set of questions that encompass three domains of food insecurity: (1) anxiety and uncertainty about the household food supply; (2) insufficient quality; and (3) insufficient food intake and its physical consequences (Coates et al. 2007).
  Each household receives a score from 0-27 based on a simple sum of the frequency of occurrence of each food insecurity condition, where 'never' = 0 points, 'rarely' = 1 point, 'sometimes' = 2 points, and 'often' = 3 points. The higher the score, the higher the degree of household food insecurity experienced in the previous four weeks.

CONTACTS AND LOCATIONS:
Overall Officials: Stefaan De Henauw, Md. PhD, Principal Investigator — University Ghent; Souheila Abbeddou, MSc. PhD, Principal Investigator — University Ghent; Hilda Vasanthakaalam, PhD, Principal Investigator — University of Rwanda; Jerome Some, Md. PhD, Principal Investigator — Institut de Recherche en Sciences de la Sante, Ouagadougou, Burkina Faso
Locations (1):
- University of Rwanda, Kigali, Rwanda

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bowen L, Ebrahim S, De Stavola B, Ness A, Kinra S, Bharathi AV, Prabhakaran D, Reddy KS. Dietary intake and rural-urban migration in India: a cross-sectional study. PLoS One. 2011;6(6):e14822. doi: 10.1371/journal.pone.0014822. Epub 2011 Jun 22. PMID 21731604
- [Background] Boutayeb A. The double burden of communicable and non-communicable diseases in developing countries. Trans R Soc Trop Med Hyg. 2006 Mar;100(3):191-9. doi: 10.1016/j.trstmh.2005.07.021. Epub 2005 Nov 4. PMID 16274715
- [Background] Swinburn BA, Kraak VI, Allender S, Atkins VJ, Baker PI, Bogard JR, Brinsden H, Calvillo A, De Schutter O, Devarajan R, Ezzati M, Friel S, Goenka S, Hammond RA, Hastings G, Hawkes C, Herrero M, Hovmand PS, Howden M, Jaacks LM, Kapetanaki AB, Kasman M, Kuhnlein HV, Kumanyika SK, Larijani B, Lobstein T, Long MW, Matsudo VKR, Mills SDH, Morgan G, Morshed A, Nece PM, Pan A, Patterson DW, Sacks G, Shekar M, Simmons GL, Smit W, Tootee A, Vandevijvere S, Waterlander WE, Wolfenden L, Dietz WH. The Global Syndemic of Obesity, Undernutrition, and Climate Change: The Lancet Commission report. Lancet. 2019 Feb 23;393(10173):791-846. doi: 10.1016/S0140-6736(18)32822-8. Epub 2019 Jan 27. No abstract available. PMID 30700377
- [Background] Janjua NZ, Mahmood B, Bhatti JA, Khan MI. Association of household and community socioeconomic position and urbanicity with underweight and overweight among women in Pakistan. PLoS One. 2015 Apr 2;10(4):e0122314. doi: 10.1371/journal.pone.0122314. eCollection 2015. PMID 25835540